CLINICAL TRIAL: NCT00691522
Title: Open-Label, Imaging Study of Human Corticotropin-Releasing Factor (hCRF) for The Reduction of Peritumoral Brain Edema (PBE) in Patients With Primary Malignant or Metastatic Brain Tumors
Brief Title: Imaging Study of XERECEPT® Treatment for Peritumoral Brain Edema (PBE)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaNet (Industry)
Collaborators: Celtic Pharma Development Services (Industry)
Responsible Party: Pharmanet, Pharmanet
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPDS 0701
Expanded Access: Available
Record Dates: First submitted 2008-06-02; First posted 2008-06-05 (Estimated); Last update posted 2009-01-09 (Estimated); Status verified 2009-01

CONDITIONS: Peritumoral Brain Edema; PRIMARY MALIGNANT and METASTATIC BRAIN TUMORS
Keywords: PERITUMORAL BRAIN EDEMA; PRIMARY MALIGNANT BRAIN TUMORS; METASTATIC BRAIN TUMORS
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Xerecept

SUMMARY:
This is a phase II, multicenter, open-label, imaging study of hCRF in the reduction of PBE in patients with primary malignant or metastatic brain tumors. Approximately 30 to 60 patients will be assigned to 1 of 3 treatment groups and receive study drug for up to 28 days

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effect of 3 different regimens of subcutaneous (SC) administered hCRF (1.0 mg every [Q] 8 hours [h], 1.5 mg Q12h, and 1.0 mg Q12h) on the reduction of PBE in patients with primary malignant or metastatic brain tumors as defined by MRI indexes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Written informed consent has been provided and documented.
* Primary malignant or metastatic brain tumor that is either asymptomatic or symptomatic patients with the life expectancy estimation of 3 months or more
* A pretreatment MRI brain scan must identify at least 1 dominant tumor lesion and related PBE that is radiologically (or visibly) distinct from the main tumor mass; the combined tumor-edema lesion must be > 2 cm in longest diameter (for at least 1 slice) and visible in 3 consecutive, 4 mm sections on MRI.
* No dexamethasone or anti-angiogenic treatment for at least 14 days prior to the Baseline and throughout the study.
* A Karnofsky Performance Score > 60 at Screening (Visit 1) and at Baseline
* A negative serum pregnancy test at the Screening (Visit 1) is required for women of childbearing potential.

Exclusion Criteria:

* • Low-grade gliomas, recurrent gliomas, suspected lymphoma, or known human immunosuppressive virus (HIV) infection.

  * Patients requiring surgery, radiosurgery or radiation surgery therapy
  * Patients experiencing severe symptoms related to PBE
  * Patients where MRI is contraindicated for any reason.
  * Signs and/or symptoms of relatively severe cerebral herniation.
  * Concurrent enrollment in any other investigational drug or device study, or plan to enroll in such a study during the 3 to 4 weeks of study treatment.
  * Systemic corticosteroid use (with the exception of inhalers for asthma).
  * Use of dexamethasone (eg, as an anti-emetic) during screening or during the study
  * Use of anti-angiogenic/anti-vascular endothelial growth factor (VEGF) therapy or anticonvulsant therapy (if patient's liver function tests (LFTs) are > 3 times upper limit of normal) 14 days prior to randomization
  * Serious concomitant cardiovascular, pulmonary, renal, gastrointestinal, or endocrine metabolic disease, which in the opinion of the Investigator or the Medical Monitor, would put the patient as unusual risk during study participation.
  * Known renal insufficiency or screening glomerular filtration rate (GFR) < 60 mL/min/1.73 m2.
  * Central nervous system infection, human immunosuppressive virus (HIV) positive or ongoing infectious process.
  * For female patients: pregnancy, breastfeeding or refusal to practice birth control if of childbearing potential during the study.
  * Inability of the patient to follow the treatment regimen.
  * Known history of methionine allergy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-08 (Estimated); Study Completion 2009-10 (Estimated)